CLINICAL TRIAL: NCT03555916
Title: Use of Botulinum Toxin (BTX) for the Treatment of Peripheral Painful Traumatic Trigeminal Neuropathy (PPTTN)
Brief Title: Botulinum Toxin Injections for Oral Neuropathic Pain
Acronym: TRIGTOX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Karolinska Institutet (Other); University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P150901; 2017-002353-11 (EudraCT Number)
Record Dates: First submitted 2018-04-09; First posted 2018-06-14 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Trigeminal Neuropathy, Traumatic
Keywords: BOTOX®-Allergan; PPTTN; Pain measurements
MeSH Terms: conditions — Trigeminal Nerve Injuries | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug (Experimental): BOTOX®, Allergan treatment in 2 mL of saline solution (0.9% NaCl) treatment
  Interventions: Drug: BOTOX®, Allergan
- Placebo (Placebo Comparator): 2 mL of saline solution (0.9% NaCl) treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BOTOX®, Allergan — 50 U BTX-A (BOTOX®, Allergan) powder diluted in 2 mL saline solution (0.9% NaCl) administrated at visit 2 by intra oral injection
  Other Names: BOTOX
  Arms: Drug
Drug: Placebo — 2 mL saline solution (0.9% NaCl) administrated at visit 2 by intra oral injection
  Arms: Placebo

SUMMARY:
Peripheral painful traumatic trigeminal neuropathy (PPTTN) are poorly relieved by existing treatments which in addition induce many adverse effects. BTX, which blocks the exocytosis of neurotransmitters, can be captured by axonal retrograde transport in primary nociceptive neurons. Injected in the painful area, it might therefore inhibit the release of algogenic neurotransmitters, at both the peripheral and central levels and thus reduce pain. One study reported such an effect in neuropathic spinal pain. A recent study reported an analgesic effect in trigeminal neuralgia.

DETAILED DESCRIPTION:
Traumas of either physical (shocks, ballistic impacts etc.) or surgical origin are accompanied by acute pain which disappears in most cases with tissue healing. However, in some instances pain may persist in spite of an apparently normal tissue repair. Many reports have pointed to the societal impact of these neuropathic pains which is a major public health problem in Europe and in the world. In addition to the degradation of the quality of individual life that affects hedonistic, emotional, social, professional etc. dimensions of life, the economic cost to society is considerable (treatment costs, work absenteeism, loss of motivation and concentration, etc.) Among these pains, PPTTN resulting from orofacial nerve damage after physical or surgical trauma are little studied. Some studies suggest a high prevalence, ranging from 0.5 to 12% after oral surgery, including endodontic treatment (root canal treatment), simple or complex dental extractions like wisdom teeth, dental implants, and surgical interventions (cyst removal, orthognathic surgery etc.). However, despite significant advances in recent decades, pathophysiological mechanisms of these pains are still largely unknown. The majority of these pains are clinically resistant to standard analgesics and therefore extremely difficult to treat, particularly for trigeminal pain. Understanding these pains is of major interest to determine new strategies and therapeutic targets.

Symptomatology and Pathophysiology The main complaint of patients is moderate to severe and usually burning but may be stabbing. Most cases are continuous, but may report superimposed paroxysmal pain attacks. Less frequently, the pain may be short lasting with associated mechanical trigger areas, mimicking trigeminal idiopathic neuralgia. However, even in these cases, the pain attacks are usually longer than those associated with trigeminal neuralgia. Pain is unilateral and may be precisely located to the dermatome of the affected nerve with demonstrable sensory dysfunction. The pain may be diffuse and spread across dermatomes, but rarely crosses the midline. Patients may complain of a feeling of swelling, foreign body, hot or cold, local redness or flushing. Non-painful but annoying dysesthesias such as itching, numbness, etc. are often present.

From a pathophysiological point of view, the development of painful symptoms after peripheral nerve injury is related to peripheral and central changes. Damaged tissue initiate peripheral changes at the injury site that result in functional changes of neuronal, glial and vascular cells, followed by ganglionic and central changes. These changes modify both the functioning and the excitability of individual neurons and the configuration of synaptic networks, at the spinal cord/ brainstem and brain levels. These events in turn lead to genetic and epigenetic changes which translate as long term alterations of neuronal phenotypes Our research group (Team "Neuroinflammation Pain and Stress", U894, Psychiatry Centre and Neurosciences.) has been involved for many years in deciphering the actors and events contributing to the development of post-traumatic neuropathic pain, in both spinal and trigeminal models.

Treatment The diagnostic difficulty is a therapeutic challenge. During the many consultations (average of 7.5 practitioners visited), patients received different treatments: surgical, antidepressant, analgesic or alternative which are often ineffective and potentially iatrogenic and often need to be complemented by a psychotherapeutic approach.

The surgical management of patients with neuropathic pain is controversial. Indeed, the long term results of micro-neurosurgical procedures are often anecdotal, highly variable, and operator-dependent. In addition they are difficult to assess because studies are rare and involve only few patients. A thorough evaluation of these techniques is necessary and many other authors recommend stopping any surgical procedure at the site of pain and contraindicate surgery. These could indeed worsen the patient's pain.

Pharmacological treatment of PPTTN is the same as for post traumatic spinal neuropathic pain. It is symptomatic, not curative, and combines systemic medical treatment with topical treatment (anesthetics). Neuropathic pain responds little or not at all to the classical analgesics like acetaminophen or nonsteroidal anti-inflammatory drugs (NSAIDs) and are treated by other therapeutic classes. Current treatments are based on the recommendations of different scientific societies, French (SFETD), European (EFNS) and American (APS). Treatments usually used are tricyclic antidepressants, anticonvulsants, opioids and inhibitors of the reuptake of serotonin and norepinephrine. However these treatments induce many adverse effects more or less tolerated, sometimes leading to treatment discontinuation or dose reductions and impaired efficiency.

In conclusion, the diagnosis of PPTTN is difficult and is often made after extensive consultations in specialized centers. The management is unsatisfactory due to the complexity of physio-pathogenic mechanisms and the lack of specific drugs. It is most often performed by specialized practitioners and uses multidisciplinary skills (dentist, neurologist, psychiatrist and psychologist).

Hypothesis for the study Since its introduction in the 1970s for the treatment of strabismus, blepharospasm, and focal dystonia, botulinum toxin type A (BTX-A) has been widely used in the treatment of conditions characterized by excessive muscle contraction and/or involvement of the cholinergic system (focal dystonia, spasticity, abnormal sphincter contractions, eye movement, hyperkinetic and vegetative disorders). Many studies have also been conducted in the case of painful conditions with a muscular component following a pioneer work observing a significant decrease in pain after BTX injection. Other studies have also reported pain relief during several weeks. The neurotoxin has been used in other types of pain disorders including myofascial pain, blepharospasm, myalgia of the masticatory system (TMD), back pain, painful myoclonia, urologic, rectal or pelvic pain and cervicogenic, neurovascular and tension type headaches, and migraine. The results depend on conditions and on the dose used.

It is at the Neuromuscular junction (NMJ) that the action of botulinum neurotoxin has been the most studied. It blocks the release of acetylcholine and causes a reversible deafferentation of the motor endplate (28 days). A first recovery occurs by sprouting and the restoration of function in the initial innervation and loss of sprouts. Full recovery is achieved in about 90 days. However, this sole effect appears insufficient to explain all of the analgesic activity of the neurotoxin, demonstrated in numerous animal studies and therapeutic clinical trials.Effects on nociceptive system The effects of the neurotoxin can also be explained by effects other than on the neuromuscular system, including the nociceptive system. BTX affects the vesicular release of neurotransmitters / neuromodulators. The analgesic effect may be explained by a peripheral action by blocking the axon reflex that releases usually neuropeptides (substance P, neurokinin A, CGRP) by small diameter type C primary afferent nerve fibers and causes the phenomena of neurogenic inflammation including vasodilation and increased vascular permeability. BTX inhibits the release of substance P and glutamate and reduces the inflammatory pain induced by formalin injection. In addition, the toxin can be captured by nerve endings and transported by retrograde and orthograde axonal transport to remote sites, at the level of primary afferents termination site for example or at other sites of neuronal interaction with glial cells or other neuronal types. BoNT can therefore inhibit the release of algogenic neurotransmitters present in nociceptive primary afferent (SP, glutamate) both peripherally and centrally. BTX also decreases the expression of TRPV1 receptors on the membrane surface of nociceptors in animals, and humans. These receptors are involved in the transduction of thermal information and their activation results in a burning sensation, which is also a frequently encountered qualitative characteristic in post-traumatic neuropathic pain. Recently it has been shown that administration of BTX decreases the expression of TRPV1 in dorsal root ganglion neurons in a diabetic model of neuropathic pain. Finally, the toxin also decreases the expression of other pain receptors such as purinergic receptors P2X3. In humans, the intradermal injection of BTX-A in healthy volunteers resulted in a marked decrease in specific and painful mechanical sensitivity without changing the tactile, non nociceptive mechanoreception, without affecting the density of cutaneous innervation.

Injected in the painful area, BTX-A might therefore inhibit the release of algogenic neurotransmitters, at both the peripheral and central levels and thus reduce pain.

The proposed study will therefore explore in a double blind randomized, with two parallel groups, BTX-A vs placebo, the analgesic effects of BTX-A in PPTTN patients.

ELIGIBILITY:
Inclusion criteria

1. Informed consent form signed
2. Adult patients, age 18 -75 y.o.
3. Medical coverage (excepted AME)
4. Understanding of all medical information
5. Subjects fulfilling diagnostic criteria for Peripheral painful traumatic trigeminal neuropathy (PPTTN)
6. Pain in one or several branches of the trigeminal nerve
7. History of surgical treatment (including endodontic treatments) in the painful area
8. Pain in the area experienced in the 3 months following the treatment
9. pain almost every day for at least 6 months
10. VAS ≥ 30 /100 mm
11. Primary painful area limited to one dental quadrant
12. Presence of at least one positive (hyperalgesia, allodynia, numbness or swelling) and/or negative (anesthesia or hypoesthesia) sign of neurological dysfunction
13. Pain cannot be attributed to another cause

Exclusion criteria

1. Patients with impaired communication
2. Pregnancy, breastfeeding or planning pregnancy within the period of the study
3. Women of childbearing potential (WOCBP), adequate method of contraception within the period of the study
4. Orofacial pain other than PPTTN unless clearly identifiable TMD (arthralgia, muscle pain or disc displacement)
5. Contra-indications for BTX-A (for example diseases of the neuromuscular junction, known hypersensitivity to BTX-A etc.)
6. Known coagulation disorders
7. Major depression (score > XX HADS scale)
8. Background of drug consumption or excessive alcohol consumption (3 units of alcohol a day)
9. current legal dispute with a dental practitioner
10. Former use of BTX for esthetic purpose
11. Dysphagia
12. Aspiration pneumonitis
13. Troubles with bladder control
14. Concomitant use of analgesics with dosage modification since less one month before inclusion in the study
15. Topical applications of drugs and anesthetics which cannot be interrupted one week before visit sessions
16. Treatment with aminoglycosides in the three months preceding the selection
17. Participation to another interventional clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline of self-reported average pain intensity using 11-point numerical scale (0 = no pain; 10 = maximal pain imaginable) at one month | before and one month after injection
  Self-reported average pain intensity from each morning's record in a diary concerning the last 24 hours during one week, before and one month after injection

SECONDARY OUTCOMES:
Pain measurement with the 11-point numerical scale of the Brief Pain Inventory (BPI) | At baseline, 1, 3 and 6 months
  Pain recorded each morning in a diary (diary 2) concerning the last 24 hours, using the 11-point numerical scale (NS; 0 = no pain; 10 = maximal pain imaginable) of the Brief Pain Inventory (BPI) at 1 month, 3 months and 6 months. The least, average, and maximum pain intensity during the 7 days will be collected and compared to baseline.
Pain measurement with the neuropathic pain symptom inventory (NPSI) | At baseline, 1, 3 and 6 months
  Items of the neuropathic pain symptom inventory (NPSI) will be recorded during the last 24 hours on 11-points (0-10 points) numerical scales.
Pain measurement with Visual Analogic Scale (VAS) | At baseline, 1, 3 and 6 months
  Visual Analogic Scale (VAS) (from 0 mm [no pain relief] to 100 mm [maximal pain relief]).
Pain measurements with Clinical Global Impression - Improvement scale (CGI-I) | At baseline, 1, 3 and 6 months
  The Clinical Global Impression - Improvement scale (CGI-I) (a 7-point scale rating from very much improved to very much worse) will be used .
Areas of pain | At baseline, 1, 3 and 6 months
  The areas of main pain and referred pain will be reported directly from the patient to a soft foil, then digitized for measurement on Image J software.
Assessment of sensory deficit according to intraoral Quantitative Sensory Testing (QST) | At baseline, 1 month
  According to the conclusions of the European task force committee for intraoral quantitative sensory testing (QST), the QST is defined by :
  * Brush-induced allodynia will be evaluated stroking the skin with a standardized brush and will be considered as present if evoking a clear sensation of pain. The intensity of allodynia will be recorded on a 100 mm visual analog scale. Area of Brush-induced allodynia will be traced on a transparent plastic foil, and then digitized for measurement on Image J software.
  * Mechanical sensations (detection thresholds to non-painful stimuli) and pain thresholds will be measured with calibrated von Frey hairs (0.06-300gm) (Bioseb, France) (or electronic von Frey, Bioseb France).
  * Thermal sensations and pain thresholds (in °C) will be assessed with a thermoalgometer (TSA II; Medoc, Israel) with an intraoral thermode by the method of limits, with baseline temperatures adjusted to the patient's skin temperature .
Emotional state with Hospital Anxiety and Depression Scale (HADS) | At baseline, 1, 3 and 6 months
  Emotional state using the Hospital Anxiety and Depression Scale (HADS) including 14 items scored as anxiety and depression scores (each on 21)
Emotional state with Brief Pain Inventory (BPI). | At baseline, 1, 3 and 6 months
  Emotional state using items of the Brief Pain Inventory (BPI).
Movement and function | At baseline, 1, 3 and 6 months
  Interference with oral function will be measured with the Brief Pain Inventory (BPI) (with the exclusion of the item "ability to walk" changed for "ability to chew" judged more relevant here) rated from 0 (does not interfere) to 10 (complete interference).
Quality of life with Geriatric Oral Health Assessment Index (GOHAI) | At baseline, 1, 3 and 6 months
  Quality of life will be assessed with specific questionnaires Geriatric Oral Health Assessment Index (GOHAI)
Quality of life with Oral Health Impact Profile (OHIP) | At baseline, 1, 3 and 6 months
  Quality of life will be assessed with specific Oral Health Impact Profile (OHIP)
Quality of life with items of Brief Pain Inventory (BPI). | At baseline, 1, 3 and 6 months
Incidence of BTX-A - Emergent Adverse event | At baseline, 1, 3 and 6 months
  Safety of BTX-A, particularly for potential systemic adverse effects, will be assessed throughout the study. Adverse events will be declared in the case report form (CRF).
Pain related to injections of BTX-A | At baseline, 1, 3 and 6 months
  Pain related to injections will be rated as mild, moderate, or severe.
Time course of the pain: | At baseline, 1, 3 and 6 months
  measurement of the time course of the pain throughout the day with a diary (diary 1) in which the patient reports his/her pain every hour on a numeric scale (0-10) during 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Yves BOUCHER, DDS,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Groupe Hospitalier Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moreau N, Dieb W, Descroix V, Svensson P, Ernberg M, Boucher Y. Topical Review: Potential Use of Botulinum Toxin in the Management of Painful Posttraumatic Trigeminal Neuropathy. J Oral Facial Pain Headache. 2017 Winter;31(1):7-18. doi: 10.11607/ofph.1753. PMID 28118416